CLINICAL TRIAL: NCT01006993
Title: Feasibility and Safety of NeuroFlo in Stroke Patients Receiving tPA
Brief Title: Feasibility and Safety of NeuroFlo in Stroke Patients Receiving Tissue Plasminogen Activator
Acronym: FASTFlo tPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CoAxia (Industry)
Responsible Party: Lori Austin, CoAxia, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0258
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeuroFlo Treatment (Experimental)
  Interventions: Device: NeuroFlo catheter

INTERVENTIONS:
Device: NeuroFlo catheter — NeuroFlo™ catheter 45 minute treatment

SUMMARY:
To assess the safety and feasibility of using the NeuroFlo catheter to treat acute ischemic stroke patients following administration of intravenous tPA.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* NIHSS between 5-22
* Persistent clinical deficits following administration of rt-PA

Exclusion Criteria:

* Planned thrombectomy
* Aortic pathology
* Severe heart disease
* Other conditions the doctor will assess

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
An assessment of serious adverse events occurring in ischemic stroke patients undergoing NeuroFlo treatment. | Baseline to 30 days post-treatment

SECONDARY OUTCOMES:
Potential patient benefit will be assessed through collection of neurological indices. | Baseline through 90 days

CONTACTS AND LOCATIONS:
Overall Officials: FASTFlo Steering Committee, Study Director — Various
Locations (4):
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of Western Ontario, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
- University of Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Emery DJ, Schellinger PD, Selchen D, Douen AG, Chan R, Shuaib A, Butcher KS. Safety and feasibility of collateral blood flow augmentation after intravenous thrombolysis. Stroke. 2011 Apr;42(4):1135-7. doi: 10.1161/STROKEAHA.110.607846. Epub 2011 Feb 24. PMID 21350210